CLINICAL TRIAL: NCT01258816
Title: A Phase I Study of the Human Pharmacokinetics and Cardiac Safety of Elacytarabine
Brief Title: The Pharmacokinetics and Cardiac Properties of Elacytarabine (CP-4055)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Collaborators: Theradex (Industry); Syneos Health (Other); CardiaBase (Other); Learn & Confirm (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-109
Record Dates: First submitted 2010-11-26; First posted 2010-12-13 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Relapsed/Refractory AML
Keywords: Acute Myeloid Leukaemia (AML); Pharmacokinetics; Elacytarabine; CP-4055
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 5'-oleoyl cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Elacytarabine for infusion — Elacytarabine 2000 mg/m2/d will be administered as a continuous intravenous infusion (CIV) in a d 1-5 q3w schedule.
  Other Names: CP-4055

SUMMARY:
The purpose of the study is to investigate the pharmacokinetics (PK) and cardiac properties of elacytarabine in patients with relapsed or refractory Acute Myeloid Leukaemia (AML). The efficacy and tolerability of elacytarabine will also be assessed.

DETAILED DESCRIPTION:
Elacytarabine is an investigational drug which is not commercially available. It consists of a fatty acid that is connected to cytarabine which is commonly used in treatment of AML. Due to the connection to a fatty acid, elacytarabine might have an increased uptake in blast cells and thereby increased efficacy.

The characterisation of the pharmacokinetics of an investigational drug, as well as the cardiac safety are essential. The PK of both elacytarabine and its metabolites will be assessed at defined timepoints before, during and after infusion. The cardiac safety of elacytarabine will be evaluated by triplicate ECG recordings at the same time points as the PK assessments.

Elacytarabine will be given as a continuous infusion for 5 days. The patients may continue with further courses of elacytarabine as long as the patient benefits from treatment with elacytarabine.

ELIGIBILITY:
Inclusion¨Criteria:

1. Patients must have relapsed / refractory AML according to WHO classification (excluding acute promyelocytic leukaemia)
2. Patients must have ECOG Performance Status (PS) of 0 - 2
3. Patients must be 18 years of age or older
4. Women of child-bearing potential must have a negative serum or urine pregnancy test within two weeks prior to treatment start
5. Male and female fertile patients must use adequate contraception for the duration of the study, and males also for 3 months after the last elacytarabine dose
6. Patients must be capable of understanding and complying with protocol requirements, and they must be able and willing to sign a written informed consent

Exclusion Criteria:

1. A history of allergic reactions to egg. A history of CTCAE grade 3 or 4 allergic reactions to ara-C of
2. A history of cancer that according to the investigator might confound the assessment of the endpoints of the clinical study
3. Known positive status for human immunodeficiency virus (HIV)
4. Pregnant and nursing patients
5. Uncontrolled inter-current illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that will limit compliance with study requirements
6. Impairment of hepatic or renal function to such an extent that the patient, in the opinion of the investigator, will be exposed to an excessive risk if entered into the clinical study
7. Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medications, or uncontrolled congestive heart failure. Any NYHA grade 3 or 4
8. A history of familial long QT syndrome
9. Patients with history of serious ventricular arrhythmia (VT or VT)
10. ECG criteria at the eligibility visit: QTc ≥ 480 msec calculated using Fridericia's correction (QTcF = QT/RRO,33) or bradycardia (<50bpm) or criteria for left ventricular hypertrophy
11. treatment with any medications known to produce QT prolongations
12. Treatment with hydroxyurea or 6-mercaptopurine within the last 12 hours prior to treatment on this protocol or any other investigational or standard cytotoxic treatment within the last 14 days

9. Any medical condition which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Characterise the pharmacokinetics of elacytarabine in patients with relapsed/refractory Acute Myeloid Leukaemia | During first week of treatment course
  Collection of pheripheral blood samples at specified time points during first week of the treatment course for PK analyses

SECONDARY OUTCOMES:
Investigate the activity of elacytarabine measured as remission rate (CR + CRi) | After each course
  Bone marrow and/or blood examination
Number of patients with Adverse Events as a measure of safety and tolerability | Continuously during study
Evaluate the cardiac safety of elacytarabine with focus on the QT/QTc intervals | During the first week of treatment
  Triplicate 12-lead ECG assessments will be done at specified time points before, during and after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Steven Knapper, MD, Principal Investigator — Cardiff University
Locations (6):
- Spain (3):
  - ICO - Hospital Duran i Reynals, Barcelona, Catalonia
  - Hospital General de la Vall d' Hebron, Barcelona
  - Hospital San Pedro Alcantara, Cáceres
- United Kingdom (3):
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - University Hospital of Wales, Cardiff, Cardiff
  - St Bartholomew's Hospital, London

REFERENCES:
- [Derived] Knapper S, Chevassut T, Duarte R, Bergua JM, Salamero O, Johansen M, Jacobsen TF, Hals PA, Rasch W, Gianella-Borradori A, Smith M. Elacytarabine in relapsed/refractory acute myeloid leukaemia: an evaluation of clinical efficacy, pharmacokinetics, cardiac safety and effects on lipid profile. Leuk Res. 2014 Mar;38(3):346-51. doi: 10.1016/j.leukres.2013.12.011. Epub 2013 Dec 25. PMID 24433865